CLINICAL TRIAL: NCT04327609
Title: SAVE Trial - Use of the Selution Sirolimus Eluting Balloon for Dysfunctional AV accEss Treatment Indications
Acronym: SAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.A. Med Alliance S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEL-001-2019
Record Dates: First submitted 2020-02-20; First posted 2020-03-31 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: AV Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SELUTION SLR™ DEB (Experimental): Med Alliance SELUTION SLR™ 018 DEB Sirolimus Eluting Balloon Catheter.
  Interventions: Device: SELUTION SLR™ DEB
- Control Treatment (Active Comparator): POBA
  Interventions: Device: Control Arm

INTERVENTIONS:
Device: SELUTION SLR™ DEB — Subjects will receive standard high-pressure balloon angioplasty followed by local application of sirolimus with the SELUTION SLR™ 018 DEB (MedAlliance) of appropriate diameter and length to achieve full lesion coverage.
  Arms: SELUTION SLR™ DEB
Device: Control Arm — The control arm will receive standard high-pressure balloon angioplasty of appropriate diameter and length and no further lesion treatment.
  Arms: Control Treatment

SUMMARY:
Prospective multi-center single-blinded randomized controlled trial (RCT) investigating the safety and feasibility of the SELUTION SLR™ (Sustained Limus Release) 018 drug eluting balloon (DEB) for the treatment of failed AV fistula in renal dialysis patients. Patients will be randomised to either SELUTION SLR or POBA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years
* Patient is able and willing to provide written informed consent
* A Dialysis Access that has performed at least 1 successful dialysis session
* Stenosis >50% at the outflow vein (by visual estimation) with clinical circuit dysfunction
* Lesion of ≤7mm in diameter
* Lesion of up to the 70mm in length

Exclusion Criteria:

* Life expectancy <1year
* Lower extremity AVG
* Infected AVG
* Uncontrolled systemic infection
* Aneurysm or pseudoaneurysm in proposed target lesion
* Presence of previous CS or BMS
* ≥2 lesions present within the circuit
* Unable to perform protocol prescribed pre-dilation of the lesion
* Patient is female and is pregnant, or planning to become pregnant during the course of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Primary Patency of the treated lesion at 6 months post-intervention. | 6 months
  Primary patency: Defined as uninterrupted patency after the initial intervention with regular ongoing dialysis until symptomatic recurrent stenosis of the dialysis circuit, or thrombosis, mandating repeat treatment, or further surgical intervention of the access circuit or eventual failure/abandonment of the circuit with creation of alternative access for dialysis. This endpoint will be analysed cumulatively at 6 months and with time-to-event methods (e.g. Kaplan Meier) on extended follow-up period to 2 years.
Freedom from any serious adverse event(s) involving the AV access circuit or the patient at 30 days | 30 days
  Freedom from any serious adverse event(s) involving the AV access circuit or the patient at 30 days.

SECONDARY OUTCOMES:
Freedom from any serious adverse event(s) involving the AV access circuit or the patient at 6 months. | 6 months
  Freedom from any serious adverse event(s) involving the AV access circuit or the patient at 6 months.
Late lumen loss | 6 months
  Late lumen loss (LLL) defined as the difference between the minimum lumen diameters after angioplasty and at the end of the 6-month follow-up angiogram.
Device Success | During Procedure
  Device Success: Defined as successful balloon inflation of the SELUTION catheter for ≥2 minutes and retrieval of the catheter.
Anatomic success | Immediately after angioplasty
  Anatomic success: Defined as <30% residual stenosis diameter measured immediately after angioplasty.
Clinical Success | 6 months
  Clinical Success: Defined as an improvement from baseline in the clinical or hemodynamic parameter (e.g., blood flow, venous pressures) that was the initial indicator of fistula dysfunction and the resumption of normal hemodialysis for a minimum of at least 1 session following the procedure.
Binary Vessel Restenosis | 6 months
  Binary vessel restenosis: Angiographic restenosis rate defined as the incidence of stenosis ≥50% of the diameter of the reference vessel segment within the treated target lesion.

CONTACTS AND LOCATIONS:
Locations (3):
- Greece (2):
  - University of Athens, Athens
  - University of Patras, Pátrai
- Singapore General Hospital LTD, Singapore, Singapore